CLINICAL TRIAL: NCT05764642
Title: Renal Microvessel Imaging for Characterization of Chronic Kidney Disease
Brief Title: A Study of Renal Microvessel Imaging for Chronic Kidney Disease
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Shigao Chen, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-006499; R01DK129205 (NIH)
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Healthy; Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Chronic Kidney Disease Group (Experimental): Subjects with Chronic Kidney Disease (CKD) with clinically indicated renal biopsy will have microvessel images obtained by Super-Resolution Ultrasound Imaging (SRUI) using Definity ultrasound contrast agent.
  Interventions: Drug: Definity; Diagnostic Test: Super-resolution ultrasound imaging
- Healthy Control Group (Active Comparator): Healthy volunteers with normal eGFR will have microvessel images obtained by Super-Resolution Ultrasound Imaging (SRUI) using Definity ultrasound contrast agent.
  Interventions: Drug: Definity; Diagnostic Test: Super-resolution ultrasound imaging

INTERVENTIONS:
Drug: Definity — Ultrasound contrast agent administered intravenously
  Other Names: Perflutren Lipid Microsphere
Diagnostic Test: Super-resolution ultrasound imaging — Imaging technology for microvessel imaging. This technology localizes and tracks individual microbubbles (FDA approved ultrasound contrast agents) to map microvessel morphology and flow speed at a spatial resolution about 10 times higher than conventional ultrasound imaging.
  Other Names: SRUI

SUMMARY:
The purpose of this research is to study the efficacy of ultrasound microvessel imaging for evaluation of Chronic Kidney Disease. Definity is an ultrasound contrast agent currently approved by the FDA for use on the heart, liver, and urinary tract. This study will look at its effectiveness on the kidney.

ELIGIBILITY:
Inclusion Criteria:

- Healthy volunteers or Chronic Kidney Disease (CKD) patients with clinically indicated renal biopsy.

Exclusion Criteria:

* Subjects lacking capacity to consent.
* Vulnerable subjects such as prisoners; pregnant women; nursing mother.
* Subjects with history of hypersensitivity allergic reactions to ultrasound contrast agents.
* Patients with high-risk cardiac diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Renal cortex microvessel density | Baseline
  Super-Resolution Ultrasound Imaging (SRUI) parameters reported in percentage
Renal cortex microvessel diameter | Baseline
  Super-Resolution Ultrasound Imaging (SRUI) parameters reported in millimeters (mm)
Renal blood flow velocity | Baseline
  Super-Resolution Ultrasound Imaging (SRUI) parameters reported in centimeters per second (cm/sec)

CONTACTS AND LOCATIONS:
Overall Officials: Shigao Chen, PhD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic Minnesota, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No